CLINICAL TRIAL: NCT02708394
Title: Molecular Mechanisms of Antipsychotic-induced Insulin Resistance in Healthy Volunteers
Brief Title: Molecular Mechanisms of Antipsychotic-induced Insulin Resistance
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Kyle Jon Burghardt, Pharm.D., Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MMAAPWSU
Record Dates: First submitted 2016-03-05; First posted 2016-03-15 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Adverse Effect of Other Antipsychotics and Neuroleptics; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- olanzapine (Experimental): Atypical antipsychotic
  Interventions: Drug: olanzapine
- placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: olanzapine — atypical antipsychotic
  Other Names: Zyprexa
  Arms: olanzapine
Drug: placebo — placebo control
  Arms: placebo

SUMMARY:
This study will investigate the molecular mechanisms of atypical-antipsychotic induced insulin resistance. This will be accomplished by administering olanzapine or placebo to healthy subjects for 7 days and analyzing genetic and protein changes in peripheral tissues known to play an important role in insulin resistance pathophysiology.

ELIGIBILITY:
We will include persons that meet the following criteria:

1. 21-45 years old
2. BMI 18.5-24.9kg/m2
3. No history of drug or alcohol dependence or abuse
4. No current or past history of psychiatric or neurologic disease
5. minimal exercise routine prior or during study (light walking allowed)
6. Normal liver function tests
7. minimal alcohol intake (<1 drink per day).

The following persons will be excluded:

1. Has 1st degree relative with diabetes (I or II)
2. current or re-cent nicotine intake
3. presence of organic/physical disease that could affect glucose
4. currently taking prescription or over-the-counter medications that could affect glucose
5. currently pregnant or lactating
6. unwilling to take acceptable birth control method
7. current or previous exposure to antipsychotics
8. history of unstable weight
9. personal or family history of cardiac arrhythmias or seizures
10. current or past history of eating disorder(s) or restricted diet
11. allergy to lidocaine or drug excipients
12. history of difficulty with intravenous line placement
13. history of fainting.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in DNA methylation | Baseline (day 1) to endpoint of intervention (day 7)
  Change in peripheral tissue candidate gene methylation will be measured in the olanzapine intervention group compared to placebo

SECONDARY OUTCOMES:
Change in protein levels | Baseline (day 1) to endpoint of intervention (day 7)
  Change in peripheral tissue candidate protein levels will be measured in the olanzapine intervention group compared to placebo
Change in protein activity | Baseline (day 1) to endpoint of intervention (day 7)
  Change in peripheral tissue candidate protein phosphorylation will be measured in the olanzapine intervention group compared to placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University Clinical Research Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT02708394/ICF_000.pdf